CLINICAL TRIAL: NCT06643416
Title: Efficacy and Safety of Add-on Topical Timolol in the Management of Epidermal Growth Factor and Anaplastic Lymphoma Kinase Receptor Tyrosine Kinase Inhibitor-induced Paronychia: a Prospective Randomized Open-labelled Trial
Brief Title: Efficacy and Safety of Add-on Timolol for EGFR-TKI and ALK-TKI Induced Paronychia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Wang Chun, Clinical Assistant Professor, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-573
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Paronychia; EGFR-TKI; ALK-TKI
Keywords: EGFR TKI; paronychia; timolol; ALK-TKI
MeSH Terms: conditions — Paronychia | interventions — Timolol; Ophthalmic Solutions; Betamethasone Valerate

STUDY DESIGN:
Intervention Model Description: 40 Adult patients aged 18 or above who received EGFR-TKI and ALK-TKI, namely gefitinib, erlotinib, afatinib, osimertinib, amivantamab, dacomitinib, mobocertinib, crizotinib, ceritinib, alectinib, brigatinib and lorlatinib for the treatment of non-small cell lung cancer, who develop paronychia (affecting fingernails, toenails or both),as an adverse event from EGFR-TKI use will be included in this study. Patients will be randomized in 1:1 ratio using computer-generated randomization list to receive either combination of topical timolol 0.5% eye drops and betamethasone valerate 0.1% lotion application twice daily or betamethasone valerate 0.1% lotion application twice daily.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Timolol combination treatment (Active Comparator): Patients will received topical timolol 0.5% eye drops (liquid form) twice daily with occlusion (i.e. covered with adhesive badge) and betamethasone valerate 0.1% cream twice daily with occlsuion for 1 month. For patients who do not have paronychia completely resolved after 4 weeks, the treatment assigned will be continued for another 4 to 8 weeks, up to 12 weeks to see the effect.
  Interventions: Drug: Timolol 0.5% eye drops and betamethasone valerate 0.1% cream; Drug: Betamethasone valerate 0.1% cream
- Routine Arm (Other): Patients in routine arm would receive the management according to routine clinical practice, including prescription of betamethasone valerate 0.1% cream twice daily for 1 month with occlusion. For patients who do not have paronychia completely resolved after 4 weeks, the treatment assigned will be continued for another 4 to 8 weeks, up to 12 weeks to see the effect.
  Interventions: Drug: Betamethasone valerate 0.1% cream

INTERVENTIONS:
Drug: Timolol 0.5% eye drops and betamethasone valerate 0.1% cream — Topical timolol 0.5% eye drops (liquid form) twice daily with occlusion (i.e. covered with adhesive badge) and betamethasone valerate 0.1% cream twice daily with occlsuion for 1 month. For patients who do not have paronychia completely resolved after 4 weeks, the treatment assigned will be continued for another 4 to 8 weeks, up to 12 weeks to see the effect.
  Arms: Timolol combination treatment
Drug: Betamethasone valerate 0.1% cream — The management according to routine clinical practice, including prescription of betamethasone valerate 0.1% cream twice daily for 1 month with occlusion. For patients who do not have paronychia completely resolved after 4 weeks, the treatment assigned will be continued for another 4 to 8 weeks, up to 12 weeks to see the effect.

SUMMARY:
To assess the clinical efficacy of add-on topical timolol 0.5% eye drops to betamethasone valerate 0.1% for the treatment of EGFR-TKI and ALK-TKI induced paronychia.

DETAILED DESCRIPTION:
Lung cancer is the second leading cause of cancer and the leading cause of cancer-related death in Hong Kong. Non-small cell lung cancer (NSCLC) accounts for 85% of lung cancer patients. Adenocarcinoma and squamous cell carcinoma accounts for 40% and 25-30% of NSCLC patients, respectively. More than 75% of patients are diagnosed with stage III and IV lung cancer. The age-standardized one-year overall survival rate of stage III and IV NSCLC are 35-46% and 15.9-15.6%, respectively. Therefore, the management of locally advanced and metastatic lung cancer is important to improve the overall survival of NSCLC patients.

The management of locally advanced and metastatic NSCLC is actionable driver mutation dependent. Patients are recommended to have tissue biopsy to detect the actionable driver mutation. Epidermal growth factor receptor (EGFR) mutation accounts for 55.4% of actionable driver mutation in Hong Kong. Patients with EGFR mutation positive are recommended to receive EGFR tyrosine kinase inhibitor (EGFR-TKI) by the European Society of Medical Oncology and the National Comprehensive Cancer Network. Anaplastic lymphoma kinase (ALK) is another common is actionable driver mutation with tyrosine kinase inhibitor (TKI) including crizotinib, ceritinib, alectinib, brigatinib and lorlatinib.

Paronychia is one of the common adverse events in patients who receive EGFR-TKI(s) and other TKI. 17.6-57% of patients experienced paronychia in randomized controlled trials. There were 0.6-11% of patients who experienced grade 3 paronychia according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAEv5.0) in randomized controlled trials.

Timolol and betaxolol are beta-blockers, which are hypothesized to be effective in managing paronychia. Beta-blockers were effective in hemangiomas and has been the first line treatment for severe infantile hemangiomas. Previous case reports and case series suggested the potential use of topical beta-blocker. However, the evidence of topical beta-blocker treatment was limited by small sample size and low level of evidence. Therefore, this study aims to compare the safety and efficacy of topical timolol with routine clinical care with paronychia (fingernails, toenails, or both) as an adverse effect of EGFR-TKI and ALK-TKI.

This study would assess the clinical efficacy of add-on topical timolol 0.5% eye drops to betamethasone valerate 0.1% for the treatment of EGFR-TKI and ALK-TKI induced paronychia. Eligible patients, who develop paronychia (affecting fingernails, toenails or both), will be included in this study. They will be randomized in 1:1 ratio using computer-generated randomization list to receive either combination of topical timolol 0.5% eye drops and betamethasone valerate 0.1% lotion application twice daily or betamethasone valerate 0.1% lotion application twice daily. Patients in timolol combination treatment group will receive topical timolol 0.5% eye drops twice daily with occlusion (i.e. covered with adhesive badge) and betamethasone valerate 0.1% lotion twice daily with occlusion for 1 month. Patients in routine arm would receive the management according to routine clinical practice, including prescription of betamethasone valerate 0.1% lotion twice daily for 1 month with occlusion. For patients who do not have paronychia completely resolved after 4 weeks, the treatment assigned will be continued for another 4 to 8 weeks , up to 12 weeks to see the effect.

ELIGIBILITY:
Inclusion criteria

1. Aged 18 years or above, either males or females.
2. Received EGFR-TKI and ALK-TKI, namely gefitinib, erlotinib, afatinib, osimertinib, amivantamab, dacomitinib, mobocertinib, crizotinib, ceritinib, alectinib, brigatinib and lorlatinib for the treatment of non-small cell lung cancer.
3. Paronychia (fingernails, toenails, or both) as an adverse event from EGFR-TKI use
4. Written informed consent obtained from patient
5. Subjects are diagnosed with advanced non-small cell lung cancer

Exclusion criteria

1. 1. Age below18
2. 2. Patients who are allergic to, or contraindicated to topical timolol use
3. 3. Pregnant women or nursing mother
4. 4. Non-consenting patients
5. 5. Subjects are not diagnosed with advanced non-small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieved complete response (disappearance of the lesion, absent pain, and/or bleeding) on topical timolol 0.5% eye drops as compared to betamethasone valerate 0.1% lotion | From baseline to month 3
  The proportion of patients achieved complete response (disappearance of the lesion, absent pain, and/or bleeding) on topical timolol 0.5% eye drops as compared to betamethasone valerate 0.1% lotion

SECONDARY OUTCOMES:
The proportion of patients achieved complete or partial response | From baseline to month 3
  Proportion of patients achieved complete or partial response (improvement in at least 1 of these 3 items).
Lack of response as well as proportion of patients with reduced severity of paronychia | From baseline to month 3
  Proportion of patients lack of response (improvement in less than 1 item)
Change in chronic paronychia severity index scale with treatment | From baseline to month 3
  Involvement of 1 nail fold = 1; involvement of 2 nail folds [proximal or/and lateral] = 2; bilateral lateral nail fold involvement and proximal nail fold involvement = 3), edema (absent = 0; mild = 1; moderate = 2; severe = 3), erythema (absent = 0; mild = 1; moderate = 2; severe = 3), nail plate changes (absent = 0; mild = 1; moderate = 2; severe = 3), and cuticle involvement (normal = 0; damaged = 1; absent = 2), producing a combined total score (between 0 [min.] and 14 [max.]
The improvement of paronychia by 4 point scale | From baseline to month 3
  1: 0 to <30%, 2: 30 to <50%, 3: 50 to 75%, 4: 75 to 100% improvement
Change in severity of pain by Visual Analog Scale | From baseline to month 3
  VAS scores ≤3.4cm corresponded to mild pain-related interference with functioning, scores of 3.5-6.4 to moderate interference, and scores ≥6.5 to severe interference.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
privacy and confidentiality

REFERENCES:
- [Background] Atis G, Goktay F, Altan Ferhatoglu Z, Kaynak E, Sevim Kecici A, Yasar S, Aytekin S. A Proposal for a New Severity Index for the Evaluation of Chronic Paronychia. Skin Appendage Disord. 2018 Nov;5(1):32-37. doi: 10.1159/000489024. Epub 2018 May 30. PMID 30643778
- [Background] Martinez-de-Espronceda I, Bernabeu-Wittel J, Azcona M, Monserrat MT. Recalcitrant trametinib-induced paronychia treated successfully with topical timolol in a pediatric patient. Dermatol Ther. 2020 Jan;33(1):e13164. doi: 10.1111/dth.13164. Epub 2019 Nov 15. PMID 31705590
- [Background] Sibaud V, Casassa E, D'Andrea M. Are topical beta-blockers really effective "in real life" for targeted therapy-induced paronychia. Support Care Cancer. 2019 Jul;27(7):2341-2343. doi: 10.1007/s00520-019-04690-8. Epub 2019 Mar 7. PMID 30847700
- [Background] Walters S, Maringe C, Coleman MP, Peake MD, Butler J, Young N, Bergstrom S, Hanna L, Jakobsen E, Kolbeck K, Sundstrom S, Engholm G, Gavin A, Gjerstorff ML, Hatcher J, Johannesen TB, Linklater KM, McGahan CE, Steward J, Tracey E, Turner D, Richards MA, Rachet B; ICBP Module 1 Working Group. Lung cancer survival and stage at diagnosis in Australia, Canada, Denmark, Norway, Sweden and the UK: a population-based study, 2004-2007. Thorax. 2013 Jun;68(6):551-64. doi: 10.1136/thoraxjnl-2012-202297. Epub 2013 Feb 11. PMID 23399908
- [Background] Puttgen K, Lucky A, Adams D, Pope E, McCuaig C, Powell J, Feigenbaum D, Savva Y, Baselga E, Holland K, Drolet B, Siegel D, Morel KD, Garzon MC, Mathes E, Lauren C, Nopper A, Horii K, Newell B, Song W, Frieden I; Hemangioma Investigator Group. Topical Timolol Maleate Treatment of Infantile Hemangiomas. Pediatrics. 2016 Sep;138(3):e20160355. doi: 10.1542/peds.2016-0355. Epub 2016 Aug 15. PMID 27527799
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Background] Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Lee KY, Xu CR, Massey D, Kim M, Shi Y, Geater SL. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):213-22. doi: 10.1016/S1470-2045(13)70604-1. Epub 2014 Jan 15. PMID 24439929
- [Background] Paz-Ares L, Tan EH, O'Byrne K, Zhang L, Hirsh V, Boyer M, Yang JC, Mok T, Lee KH, Lu S, Shi Y, Lee DH, Laskin J, Kim DW, Laurie SA, Kolbeck K, Fan J, Dodd N, Marten A, Park K. Afatinib versus gefitinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: overall survival data from the phase IIb LUX-Lung 7 trial. Ann Oncol. 2017 Feb 1;28(2):270-277. doi: 10.1093/annonc/mdw611. PMID 28426106
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Background] Yatabe Y, Kerr KM, Utomo A, Rajadurai P, Tran VK, Du X, Chou TY, Enriquez ML, Lee GK, Iqbal J, Shuangshoti S, Chung JH, Hagiwara K, Liang Z, Normanno N, Park K, Toyooka S, Tsai CM, Waring P, Zhang L, McCormack R, Ratcliffe M, Itoh Y, Sugeno M, Mok T. EGFR mutation testing practices within the Asia Pacific region: results of a multicenter diagnostic survey. J Thorac Oncol. 2015 Mar;10(3):438-45. doi: 10.1097/JTO.0000000000000422. PMID 25376513
- [Background] Planchard D, Popat S, Kerr K, Novello S, Smit EF, Faivre-Finn C, Mok TS, Reck M, Van Schil PE, Hellmann MD, Peters S; ESMO Guidelines Committee. Metastatic non-small cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv192-iv237. doi: 10.1093/annonc/mdy275. No abstract available. PMID 30285222
- [Background] Cubiro X, Planas-Ciudad S, Garcia-Muret MP, Puig L. Topical Timolol for Paronychia and Pseudopyogenic Granuloma in Patients Treated With Epidermal Growth Factor Receptor Inhibitors and Capecitabine. JAMA Dermatol. 2018 Jan 1;154(1):99-100. doi: 10.1001/jamadermatol.2017.4120. PMID 29117285
- [Background] Yen CF, Hsu CK, Lu CW. Topical betaxolol for treating relapsing paronychia with pyogenic granuloma-like lesions induced by epidermal growth factor receptor inhibitors. J Am Acad Dermatol. 2018 Jun;78(6):e143-e144. doi: 10.1016/j.jaad.2018.01.015. Epub 2018 Jan 12. No abstract available. PMID 29339238
- [Background] Hagen R, Ghareeb E, Jalali O, Zinn Z. Infantile hemangiomas: what have we learned from propranolol? Curr Opin Pediatr. 2018 Aug;30(4):499-504. doi: 10.1097/MOP.0000000000000650. PMID 29846253
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Duma N, Santana-Davila R, Molina JR. Non-Small Cell Lung Cancer: Epidemiology, Screening, Diagnosis, and Treatment. Mayo Clin Proc. 2019 Aug;94(8):1623-1640. doi: 10.1016/j.mayocp.2019.01.013. PMID 31378236